CLINICAL TRIAL: NCT07328321
Title: Development and Preliminary Validation of the Cancer Pathology Acceptance Questionnaire in Women With Breast Cancer
Brief Title: Development and Assessment of the 8-item Chronic Pain Acceptance Questionnaire to Measure Disease Acceptance in Women With Breast Cancer
Acronym: CPAQ-8-BC
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Principal Investigator, Associate Professor, G. d'Annunzio University
Other Study IDs: Protocol No. 53-2023
Record Dates: First submitted 2025-12-16; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Psychological Adaptation; Psychometrics
Keywords: Breast Cancer; Neoplasm; Disease Acceptance; Psychometrics; Questionnaire; Rehabilitation; Psychological Flexibility; Commitment
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women diagnosed with Breast Cancer for Psychometric Evaluation: This group consists of 101 women with a histologically confirmed diagnosis of Breast Cancer (BC). Participants were consecutively enrolled from two inpatient Hospital Breast Units in Italy. The purpose of this group was to serve as the population for the preliminary validation of the Cancer Pathology Acceptance Questionnaire for BC (CPAQ-8-BC). The group was evaluated in a cross-sectional manner, meaning data was collected at a single point in time.
  Interventions: Behavioral: Cancer Pathology Acceptance Questionnaire

INTERVENTIONS:
Behavioral: Cancer Pathology Acceptance Questionnaire — A self-reported questionnaire (CPAQ-8-BC) designed to assess two related dimensions of disease acceptance in women with breast cancer: Activity Engagement and Disease Receptivity. The instrument is used to measure psychological flexibility and experimental avoidance in this population.

SUMMARY:
This observational study was conducted to develop and test a new self-report questionnaire, the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC), specifically adapted for women diagnosed with Breast Cancer (BC). The primary goal is to evaluate if this new tool is a reliable and valid measure for assessing disease acceptance - defined as the psychological ability to acknowledge and experience cancer-related thoughts, emotions, and physical sensations without excessive avoidance or struggle. The study investigates whether the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) accurately measures two distinct aspects: the psychological receptivity to the illness (Disease Receptivity) and the commitment to activity engagement despite the disease (Activity Engagement). This short questionnaire is intended for use by healthcare providers and rehabilitation specialists to identify patients who struggle with acceptance, potentially guiding personalized psychological therapies, such as Acceptance and Commitment Therapy (ACT), and improving participation in rehabilitation and overall quality of survivorship.

DETAILED DESCRIPTION:
Study Background and Rationale Breast Cancer (BC) remains a major global health challenge that often leads to long-term psychological distress, body image concerns, and fatigue, even after the completion of medical treatment. Disease acceptance has emerged as a key determinant of positive emotional and functional outcomes. Therefore, reliable and valid instruments are necessary to quantify acceptance in the context of Breast Cancer (BC) for both research and clinical practice.

This study addresses the limited availability of disease-specific outcome measures by developing the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC). This instrument is an adaptation of the 8-item Chronic Pain Acceptance Questionnaire (CPAQ-8). The adaptation process involved replacing the words "pain" and "chronic pain" with the terms "tumor" or "disease" to make the instrument context-specific for patients.

Methodology and Participants This is a cross-sectional, observational study approved by the University Ethical Review Committee of Sapienza University of Rome (Protocol No. 53-2023).

Sample Size: A total of 101 women with a confirmed histopathological diagnosis of Breast Cancer (BC) were consecutively enrolled from two inpatient Hospital Breast Units.

Inclusion Criteria: Adult age, confirmed Breast Cancer (BC) diagnosis, and the ability to understand the Italian language.

Data Collection: Participants filled out the self-administered Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC), which consists of 8 items rated on a scale of 0 (never true) to 6 (always true). A pilot testing phase was conducted to assess the scale's face validity, appropriateness, acceptability, and feasibility.

Psychometric Evaluation Plan

The primary focus of the psychometric testing is to investigate the Structural Validity, Reliability, and Interpretability of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC):

* Structural Validity: Confirmatory Factor Analysis (CFA) is performed to test a single-factor structure against a pre-hypothesized two-factor structure consisting of Activity Engagement and Disease Receptivity. Model fit is evaluated using the Comparative Fit Index (CFI), Tucker Lewis Index (TLI), Standardized Root Mean Square Residual (SRMR), and Root Mean Square Error of Approximation (RMSEA).
* Reliability: Internal consistency is assessed using Cronbach's alpha and McDonald's omega. Test-Retest Stability is investigated using the Intraclass Correlation Coefficient (ICC2,1) over a 10-15 day period. The Standard Error of Measurement (SEM) is also calculated.
* Interpretability: The Minimum Detectable Change (MDC) is estimated to determine the smallest change in score that can be considered a true change rather than measurement error.

Clinical Relevance The Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) is intended to serve as a tool for person-oriented evaluations in multidisciplinary rehabilitation settings. Identifying patients with low acceptance levels may help clinicians identify those prone to activity avoidance and poor functional recovery. The instrument is designed to support the tailoring of interventions, such as Acceptance and Commitment Therapy (ACT) or Cognitive-Behavioral Therapy (CBT), by assessing key areas of psychological flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Adult age
* Confirmed histopathological diagnosis of Breast Cancer (BC)
* Ability to understand the Italian language

Exclusion Criteria:

* Documented peripheral or central neurological disorders
* Systemic illnesses
* Cognitive impairment
* Recent myocardial infarction
* Previous cerebrovascular events

Ages: 18 Years to 87 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is specifically focused on women who have received a diagnosis of Breast Cancer. Participation is limited to individuals who are biologically female, consistent with the typical population affected by this condition.
Study Population: The study participants were consecutively enrolled from two specific inpatient Hospital Breast Units in Italy. The population consists of women attending these units who had received a confirmed histopathological diagnosis of Breast Cancer (BC). The units served as the primary recruitment sites for the study.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Structural Validity of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) | Baseline
  This measure assesses the underlying factor structure of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC). Structural Validity is evaluated using Confirmatory Factor Analysis (CFA) to verify the hypothesized two-factor model consisting of Activity Engagement and Disease Receptivity. Success is defined by achieving predefined model fit indices, including a Comparative Fit Index (CFI) ≥ 0.90, a Tucker Lewis Index (TLI) ≥ 0.90, and a Root Mean Square Error of Approximation (RMSEA) ≤ 0.08.
  * Scale Description: The Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) is a self-administered tool consisting of 8 items.
  * Scale Scoring: Each item is rated on a 7-point Likert scale ranging from 0 ("never true") to 6 ("always true").
  * Minimum and Maximum Values: The total score ranges from a minimum of 0 to a maximum of 48.
  * Intrepretation: Higher scores indicate a higher level of disease acceptance.

SECONDARY OUTCOMES:
Reliability of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) | At enrollment (Baseline) and 10-15 days after surgery
  This measure evaluates the consistency and stability of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC). It includes the assessment of Internal Consistency for each factor (Activity Engagement and Disease Receptivity) and Test-Retest Stability.
  * Scale Description: The Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) is a self-administered questionnaire designed to quantify disease acceptance.
  * Scale Scoring: The instrument consists of 8 items, each rated on a scale of 0 ("never true") to 6 ("always true").
  * Minimum and Maximum Values: The total score ranges from a minimum of 0 to a maximum of 48.
  * Interpretation: Higher scores indicate a higher level of disease acceptance.
  * Stability Assessment: Test-Retest Stability is calculated using the Intraclass Correlation Coefficient (ICC2,1).
Interpretability of The Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) | Through study completion, an average of 15 days
  This measure determines the smallest change in the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) score that can be considered a true change rather than measurement error. This is assessed by calculating the Minimum Detectable Change (MDC) at a 95% confidence level.
  * Scale Description: The Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) is a self-administered questionnaire adapted from the 8-item Chronic Pain Acceptance Questionnaire (CPAQ-8).
  * Scale Scoring: 8 items rated on a 7-point scale (0 to 6).
  * Minimum and Maximum Values: Total scores range from 0 to 48.
  * Interpretation: Higher scores reflect greater disease acceptance. The Minimum Detectable Change (MDC) value provides the threshold for identifying clinically relevant changes in an individual patient's score.
Psychological Inflexibility measured by the Acceptance and Action Questionnaire - II (AAQ-II) | At enrollment (Baseline)
  This measure is used to establish the convergent validity of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) by assessing its association with the construct of psychological inflexibility (the opposite of psychological flexibility).
  * Scale Description: The Acceptance and Action Questionnaire - II (AAQ-II) is a widely used 7-item self-report instrument designed to measure psychological inflexibility and experiential avoidance.
  * Scale Scoring: Each item is rated on a 7-point Likert scale ranging from 1 ("never true") to 7 ("always true").
  * Minimum and Maximum Values: The total score ranges from a minimum of 7 to a maximum of 49.
  * Interpretation: Higher scores on the Acceptance and Action Questionnaire - II (AAQ-II) indicate greater levels of psychological inflexibility.
Psychological Distress measured by the Depression, Anxiety, and Stress Scale-21 (DASS-21) | At enrollment (Baseline)
  This measure is used to evaluate the concurrent validity of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) by assessing its association with general levels of psychological distress.
  * Scale Description: The Depression, Anxiety, and Stress Scale - 21 (DASS-21) is a 21-item self-report instrument designed to measure the three related negative emotional states of depression, anxiety, and tension/stress.
  * Scale Scoring: The scale consists of three subscales (7 items each). Each item is rated on a 4-point Likert scale ranging from 0 ("did not apply to me at all") to 3 ("applied to me very much or most of the time").
  * Minimum and Maximum Values: The total score for the Depression, Anxiety, and Stress Scale - 21 (DASS-21) ranges from a minimum of 0 to a maximum of 126 (or 0 to 42 for each subscale if not multiplied.
  * Interpretation: Higher scores on the Depression, Anxiety, and Stress Scale-21 (DASS-21) indicate higher levels of psychological distress.
Catastrophizing thoughts measured by the Pain Catastrophizing Scale (PCS) | At enrollment (Baseline)
  This measure is used to evaluate the convergent validity of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) by assessing its association with catastrophizing, a maladaptive cognitive-emotional response to illness or pain characterized by magnification, rumination, and helplessness.
  * Scale Description: The Pain Catastrophizing Scale (PCS) is a 13-item self-report instrument that measures three dimensions of catastrophizing: rumination, magnification, and helplessness.
  * Scale Scoring: Each item is rated on a 5-point Likert scale ranging from 0 ("not at all") to 4 ("all the time").
  * Minimum and Maximum Values: The total score ranges from a minimum of 0 to a maximum of 52.
  * Interpretation: Higher scores on the Pain Catastrophizing Scale (PCS) indicate higher levels of catastrophizing (a worse outcome).
Health-Related Quality of Life measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | At enrollment (Baseline)
  This measure is used to evaluate the concurrent validity of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) by assessing its association with the quality of life and physical, psychological, and social functioning of cancer patients.
  * Scale Scoring: Most items are rated on a 4-point Likert scale (1 = "not at all" to 4 = "very much"), except for the global health status which uses a 7-point scale. All scores are linearly transformed to a scale of 0 to 100.
  * Minimum and Maximum Values: The score for each subscale ranges from a minimum of 0 to a maximum of 100.
  Interpretation:
  For the Functional scales and the Global Health Status scale, a higher score represents a higher (better) level of functioning or quality of life.
  For the Symptom scales and items, a higher score represents a higher (worse) level of symptomatology or problems.
Breast Cancer-Specific Quality of Life measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Breast Cancer Module (EORTC QLQ-BR23) | At enrollment (Baseline)
  This measure is used to evaluate the concurrent validity of the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) by assessing its association with quality of life issues specifically related to Breast Cancer (BC), such as body image, sexual functioning, and treatment side effects.
  Scale Scoring: Items are rated on a 4-point Likert scale (1 = "not at all" to 4 = "very much"). All scores are linearly transformed to a scale of 0 to 100.
  Minimum and Maximum Values: The score for each subscale ranges from a minimum of 0 to a maximum of 100.
  Interpretation:
  For the Functional scales (e.g., Body Image), a higher score represents a higher (better) level of functioning.
  For the Symptom scales (e.g., Systemic Therapy Side Effects), a higher score represents a higher (worse) level of symptomatology or distress. It is expected that higher acceptance scores on the Cancer Pathology Acceptance Questionnaire for Breast Cancer (CPAQ-8-BC) will correlate with better functionality

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Paolucci, MD, PhD, Principal Investigator — Department of Oral, Medical Sciences and Biotechnology (DSMOB), "G. d'Annunzio" University of Chieti-Pescara
Locations (1):
- Simple Departmental Operative Unit - Breast Unit, "Santo Spirito" Hospital of Pescara, Pescara, Pescara, Italy

IPD SHARING:
Plan to Share IPD: No